CLINICAL TRIAL: NCT05285137
Title: A Phase 1, Randomized, Double-Blind, Single-Dose and Repeat Single-Dose, Dose-Escalation Study to Determine the Safety, Tolerability, and Pharmacokinetics of CD388 Intramuscular or Subcutaneous Administration in Healthy Subjects
Brief Title: Study of CD388 Intramuscular or Subcutaneous Administration in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cidara Therapeutics Inc. (Industry)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CD388.IM.SQ.1.01
Record Dates: First submitted 2022-03-08; First posted 2022-03-17 (Actual); Results first posted 2025-01-24 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- Cohort 1A (sentinel) (Experimental): Low dose level: 2 subjects randomized at a ratio of 1:1 to receive a single dose of 50 mg CD388 or placebo, administered by IM injection
  Interventions: Combination Product: CD388 Injection; Drug: Saline placebo
- Cohort 1A (main) (Experimental): Low dose level: 9 subjects randomized at a ratio of 7:2 to receive a single dose of 50 mg CD388 or placebo, administered by IM injection
  Interventions: Combination Product: CD388 Injection; Drug: Saline placebo
- Cohort 1B (sentinel) (Experimental): Low dose level: 2 subjects randomized at a ratio of 1:1 to receive a single dose of 50 mg CD388 or placebo, administered by SQ injection
  Interventions: Combination Product: CD388 Injection; Drug: Saline placebo
- Cohort 1B (main) (Experimental): Low dose level: 9 subjects randomized at a ratio of 7:2 to receive a single dose of 50 mg CD388 or placebo, administered by SQ injection
  Interventions: Combination Product: CD388 Injection; Drug: Saline placebo
- Cohort 2A (sentinel) (Experimental): Mid dose level: 2 subjects randomized at a ratio of 1:1 to receive a single dose of 150 mg CD388 or placebo, administered by IM injection, followed by another single dose of the same treatment (CD388 or placebo) administered by the same route after washout of 5 effective half-lives after the first dose
  Interventions: Combination Product: CD388 Injection; Drug: Saline placebo
- Cohort 2A (main) (Experimental): Mid dose level: 9 subjects randomized at a ratio of 7:2 to receive a single dose of 150 mg CD388 or placebo, administered by IM injection, followed by another single dose of the same treatment (CD388 or placebo) administered by the same route after washout of 5 effective half-lives after the first dose
  Interventions: Combination Product: CD388 Injection; Drug: Saline placebo
- Cohort 2B (sentinel) (Experimental): Mid dose level: 2 subjects randomized at a ratio of 1:1 to receive a single dose of 150 mg CD388 or placebo, administered by SQ injection, followed by another single dose of the same treatment (CD388 or placebo) administered by the same route after washout of 5 effective half-lives after the first dose
  Interventions: Combination Product: CD388 Injection; Drug: Saline placebo
- Cohort 2B (main) (Experimental): Mid dose level: 9 subjects randomized at a ratio of 7:2 to receive a single dose of 150 mg CD388 or placebo, administered by SQ injection, followed by another single dose of the same treatment (CD388 or placebo) administered by the same route after washout of 5 effective half-lives after the first dose
  Interventions: Combination Product: CD388 Injection; Drug: Saline placebo
- Cohort 3A (sentinel) (Experimental): High dose level: 2 subjects randomized at a ratio of 1:1 to receive a single dose of 450 mg CD388 or placebo, administered by IM injection, followed by another single dose of the same treatment (CD388 or placebo) administered by the same route after washout of 5 effective half-lives after the first dose
  Interventions: Combination Product: CD388 Injection; Drug: Saline placebo
- Cohort 3A (main) (Experimental): High dose level: 9 subjects randomized at a ratio of 7:2 to receive a single dose of 450 mg CD388 or placebo, administered by IM injection, followed by another single dose of the same treatment (CD388 or placebo) administered by the same route after washout of 5 effective half-lives after the first dose
  Interventions: Combination Product: CD388 Injection; Drug: Saline placebo
- Cohort 3B (sentinel) (Experimental): High dose level: 2 subjects randomized at a ratio of 1:1 to receive a single dose of 450 mg CD388 or placebo, administered by SQ injection, followed by another single dose of the same treatment (CD388 or placebo) administered by the same route after washout of 5 effective half-lives after the first dose
  Interventions: Combination Product: CD388 Injection; Drug: Saline placebo
- Cohort 3B (main) (Experimental): High dose level: 9 subjects randomized at a ratio of 7:2 to receive a single dose of 450 mg CD388 or placebo, administered by SQ injection, followed by another single dose of the same treatment (CD388 or placebo) administered by the same route after washout of 5 effective half-lives after the first dose
  Interventions: Combination Product: CD388 Injection; Drug: Saline placebo
- Cohort 4B (sentinel) (Experimental): Highest dose level: 2 subjects randomized at a ratio of 1:1 to receive a single dose of 900 mg CD388 or placebo, administered by SQ injection
  Interventions: Combination Product: CD388 Injection; Drug: Saline placebo
- Cohort 4B (main) (Experimental): Highest dose level: 9 subjects randomized at a ratio of 7:2 to receive a single dose of 900 mg CD388 or placebo, administered by SQ injection
  Interventions: Combination Product: CD388 Injection; Drug: Saline placebo

INTERVENTIONS:
Combination Product: CD388 Injection — CD388 liquid for injection
Drug: Saline placebo — Sterile normal saline for injection

SUMMARY:
The purpose of this first-in-human study is to determine the safety and tolerability profile of CD388 Injection, as compared to saline placebo, when administered as a single dose to healthy adult subjects by injection either in the muscle or under the skin.

DETAILED DESCRIPTION:
A Phase 1, single-center, prospective, randomized, double-blind, single-dose and repeat single-dose, dose-escalation study to determine the safety, tolerability, and pharmacokinetics of CD388 Injection, as compared to saline placebo, when dosed either by intramuscular (IM) or subcutaneous (SQ) administration to healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent.
2. Males and females 18 to 65 years of age, inclusive.
3. A female subject must meet one of the following criteria:

   1. If of childbearing potential - agrees to use a highly effective, preferably user-independent method of contraception (failure rate of <1 percent per year when used consistently and correctly) for at least 30 days prior to screening and agrees to remain on a highly effective method until 205 days after last dose of study medication. Examples of highly-effective methods of contraception include: abstinence from heterosexual intercourse; hormonal contraceptives (birth control pills, injectable/implant/insertable hormonal birth control products, transdermal patch); intrauterine device (with or without hormones); or a double barrier method (e.g., condom and spermicide).
   2. If a female of non-childbearing potential - should be surgically sterile (i.e., has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation/occlusion) or in a menopausal state (at least 1 year without menses), as confirmed by follicle-stimulating hormone (FSH) levels (≥40 milli-International units [mIU]/milliliter [mL]).
4. A woman of childbearing potential must have a negative highly sensitive serum pregnancy test (β-human chorionic gonadotropin) at screening and a negative urine pregnancy test on Day -1 before the first dose of study drug.
5. A male subject that engages in sexual activity that has the risk of pregnancy must agree to use a double barrier method (e.g., condom and spermicide) and agree to not donate sperm during the study and until at least 205 days after the last dose of the study medication.
6. Good health and without signs or symptoms of current illness.
7. Normal clinical examination, including:

   1. No physical examination findings that an Investigator determines would interfere with interpretation of study results.
   2. Screening ECG without clinically significant abnormalities.
   3. Creatinine clearance (CrCL) ≥80 mL/minute as calculated using the Cockcroft-Gault equation.
   4. Negative urine screen for drugs of abuse and alcohol at screening and Day -1.
8. Body mass index (BMI; weight in kilograms [kg] divided by height in meters [m] squared) between 18.0 and 32.0 kg/m^2, inclusive.
9. Willing to refrain from strenuous physical activity that could cause muscle aches or injury, including contact sports, at any time from screening through 30 days after any dose of study drug.
10. Subject has adequate venous access for blood collection.

Exclusion Criteria:

1. History of any hypersensitivity or allergic reaction to zanamivir or other neuraminidase inhibitors (i.e., laninamivir, oseltamivir, peramivir), or to excipients of the CD388 Injection drug formulation; or history of drug-induced exfoliative skin disorders (e.g., Stevens-Johnson syndrome [SJS], erythema multiforme, or toxic epidermal necrolysis [TEN]).
2. History of any of the following:

   1. Allergies, anaphylaxis, skin rashes (foods such as milk, eggs, medications, vaccines, polyethylene glycol [PEG], etc.).
   2. Chronic immune-mediated disease, positive first-degree family history of autoimmune diseases.
   3. Atopic dermatitis or psoriasis.
   4. Bleeding disorder.
   5. Psychiatric condition, seizures, hallucinations, anxiety, depression, or treatment for mental conditions.
   6. Migraines.
   7. Syncope, or vasovagal syndrome with injections or blood draws.
   8. Cardiac arrhythmia.
3. Subjects with one or more of the following laboratory abnormalities at screening as defined by the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events v2.1 (DAIDS 2017):

   1. Serum creatinine, Grade ≥1 (≥1.1 × upper limit of normal [ULN])
   2. Pancreatic amylase or lipase, Grade ≥2 (≥1.5 × ULN)
   3. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT), Grade ≥1 (≥1.25 × ULN)
   4. Total bilirubin, Grade ≥1 (≥1.1 × ULN)
   5. Any other toxicity Grade ≥2, except for Grade 2 elevations of triglycerides, low density lipoprotein cholesterol, and/or total cholesterol.
   6. Any other laboratory abnormality considered to be clinically significant by the Investigator.

   Note: Retesting of abnormal laboratory values that may lead to exclusion will be allowed once without prior asking approval from the Sponsor. Retesting will take place during a scheduled or unscheduled visit during screening. Subjects with a normal value at retest may be included.
4. Alcohol or drug addiction in the past 2 years.
5. Experiencing symptoms of acute illness or chronic disease within 14 days prior to check-in to the clinical research unit (CRU).
6. At screening, a positive result for hepatitis B virus surface antigen, hepatitis C virus antibody, or human immunodeficiency virus (HIV) antibody.
7. A positive result at screening or CRU check-in for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) by polymerase chain reaction (PCR). Beginning with Protocol Amendment 2, antigen testing may be used if PCR is not available.
8. Unwilling to comply with local health policy effective at the time regarding coronavirus disease 2019 (COVID-19).*
9. Women who are pregnant or nursing.
10. Received any over-the-counter (OTC) medications or nutritional supplements within 7 days, or any prescription medications within 14 days or <5 half-lives prior to dosing.
11. Current nicotine user or has quit habitual nicotine use in the 30 days prior to screening.
12. Received any vaccines or immunoglobulins within 28 days prior to dosing (90 days in case of intravenous immunoglobulin [IVIg] or biologics, or 14 days for COVID-19 vaccine).**
13. Donated blood (within 56 days of screening) or plasma (within 7 days of screening) or experienced significant blood loss or significant blood draw when participating in non-interventional clinical trials within 60 days prior to dosing.
14. Received a blood transfusion within 28 days prior to dosing.
15. Received any biologics within 90 days prior to dosing. Previous participation in another study within 30 days or 5 half-lives of the study drug, whichever is longer, prior to screening; prior participation at any time in non-invasive methodology trials in which no drugs were given is acceptable.
16. The PI considers that the volunteer should not participate in the study.

(*) Full COVID-19 vaccination prior to participation is strongly recommended.

(**) In the event a subject chooses to receive one of the two 2-dose approved or emergency-use-authorized COVID 19 vaccines (Comirnaty® [Pfizer], Spikevax™ [Moderna]) in the interval between two CRU stays (Cohort 2A/2B or Cohort 3A/3B), flexibility in timing of the second CRU stay should be applied, to allow appropriate receipt of the second vaccine dosage or booster (based on the respective vaccine label) + 14 days, to minimize risk of confounding findings/observations.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem Equils, MD, Study Director — Cidara Therapeutics Inc.; Debra J Kelsh, MD, Principal Investigator — Altasciences Clinical Kansas, Inc.
Locations (1):
- Altasciences Clinical Kansas, Inc., Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 77 participants were enrolled in the study at a single center, 33 of whom were randomized to receive study drug via intramuscular (IM) administration and 44 of whom were randomized to receive study drug via subcutaneous (SQ) administration.
Groups:
- CD388 50 mg IM: Participants randomized to receive a single dose of 50 milligrams (mg) CD388, administered by intramuscular (IM) injection.
  CD388: CD388 liquid for injection
- CD388 150 mg IM: Participants randomized to receive a single dose of 150 mg CD388, administered by IM injection, followed by another single dose of the same treatment administered by the same route after washout of 5 effective half-lives after the first dose.
  CD388: CD388 liquid for injection
- CD388 450 mg IM: Participants randomized to receive a single dose of 450 mg CD388, administered by IM injection, followed by another single dose of the same treatment administered by the same route after washout of 5 effective half-lives after the first dose.
  CD388: CD388 liquid for injection
- Pooled Placebo IM: Participants randomized to receive a single dose of saline placebo, administered by IM injection. Of these participants, those that advanced through the study in cohorts with participants in the CD388 150 mg IM and CD388 450 mg IM arms received another single dose of saline placebo administered by the same route after washout of 5 effective half-lives after the first dose.
  Saline placebo: Sterile normal saline for injection
- CD388 50 mg SQ: Participants randomized to receive a single dose of 50 mg CD388, administered by subcutaneous (SQ) injection.
  CD388: CD388 liquid for injection
- CD388 150 mg SQ: Participants randomized to receive a single dose of 150 mg CD388, administered by SQ injection, followed by another single dose of the same treatment administered by the same route after washout of 5 effective half-lives after the first dose.
  CD388: CD388 liquid for injection
- CD388 450 mg SQ: Participants randomized to receive a single dose of 450 mg CD388, administered by SQ injection, followed by another single dose of the same treatment administered by the same route after washout of 5 effective half-lives after the first dose.
  CD388: CD388 liquid for injection
- CD388 900 mg SQ: Participants randomized to receive a single dose of 900 mg CD388, administered by SQ injection.
  CD388: CD388 liquid for injection
- Pooled Placebo SQ: Participants randomized to receive a single dose of saline placebo, administered by SQ injection. Of these participants, those that advanced through the study in cohorts with participants in the CD388 150 mg SQ and CD388 450 mg SQ arms received another single dose of saline placebo administered by the same route after washout of 5 effective half-lives after the first dose.
  Saline placebo: Sterile normal saline for injection
Period: Overall Study
Arm/Group | CD388 50 mg IM | CD388 150 mg IM | CD388 450 mg IM | Pooled Placebo IM | CD388 50 mg SQ | CD388 150 mg SQ | CD388 450 mg SQ | CD388 900 mg SQ | Pooled Placebo SQ
Started | 8 | 8 | 8 | 9 | 8 | 8 | 8 | 8 | 12
Completed | 8 | 6 | 5 | 5 | 8 | 8 | 4 | 8 | 10
Not Completed | 0 | 2 | 3 | 4 | 0 | 0 | 4 | 0 | 2
Not completed — Failure to Meet Continuation Criteria | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Population included all randomized participants who received any amount of study drug (77 total; 33 [IM route], 44 [SQ route]).
Groups:
- Total: Total of all reporting groups
Arm/Group | CD388 50 mg IM | CD388 150 mg IM | CD388 450 mg IM | Pooled Placebo IM | CD388 50 mg SQ | CD388 150 mg SQ | CD388 450 mg SQ | CD388 900 mg SQ | Pooled Placebo SQ | Total
Number analyzed (Participants) | 8 | 8 | 8 | 9 | 8 | 8 | 8 | 8 | 12 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (7.77) | 41.1 (12.83) | 38.6 (12.73) | 39.0 (15.51) | 42.8 (12.58) | 32.8 (10.75) | 39.3 (14.95) | 41.9 (13.97) | 39.4 (13.82) | 39.3 (12.62)
Age, Continuous [Median (Full Range); unit: years] | 37.0 [30 to 55] | 38.5 [24 to 57] | 32.5 [28 to 63] | 30.0 [23 to 65] | 45.5 [21 to 56] | 30.5 [22 to 50] | 35.5 [19 to 62] | 34.0 [29 to 65] | 37.5 [18 to 59] | 35.0 [18 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 1 | 5 | 3 | 1 | 2 | 1 | 5 | 23
  Male | 7 | 4 | 7 | 4 | 5 | 7 | 6 | 7 | 7 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 6
  Not Hispanic or Latino | 8 | 5 | 7 | 9 | 8 | 7 | 7 | 8 | 12 | 71
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 3 | 4 | 4 | 6 | 5 | 7 | 8 | 43
  White | 5 | 4 | 4 | 3 | 4 | 2 | 3 | 1 | 4 | 30
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 86.19 (5.680) | 79.53 (11.945) | 79.51 (16.157) | 79.97 (12.596) | 83.15 (19.835) | 81.03 (17.053) | 85.28 (16.085) | 86.30 (10.079) | 76.73 (13.775) | 81.67 (13.847)
Weight [Median (Full Range); unit: kg] | 85.50 [77.6 to 95.3] | 80.40 [64.8 to 99.9] | 75.60 [63.0 to 105.9] | 80.90 [55.0 to 95.2] | 78.75 [59.9 to 112.5] | 78.20 [59.5 to 115.8] | 83.75 [64.1 to 118.6] | 87.90 [68.5 to 99.9] | 79.50 [55.4 to 101.7] | 81.70 [55.0 to 118.6]
Height [Mean (Standard Deviation); unit: centimeters] | 178.88 (8.919) | 172.25 (11.498) | 174.50 (6.655) | 172.00 (10.283) | 173.38 (11.975) | 172.38 (10.993) | 172.00 (11.514) | 176.19 (7.348) | 171.17 (7.884) | 173.49 (9.529)
Height [Median (Full Range); unit: centimeters] | 179.00 [168.0 to 193.0] | 173.50 [154.0 to 185.0] | 176.00 [164.0 to 184.0] | 177.00 [153.0 to 184.0] | 176.50 [157.0 to 190.0] | 174.00 [155.0 to 191.0] | 169.50 [159.0 to 193.0] | 176.75 [165.0 to 187.0] | 171.50 [159.0 to 186.0] | 175.00 [153.0 to 193.0]
Body Mass Index [Mean (Standard Deviation); unit: kilograms/meter^2 (kg/m^2)] | 27.10 (3.033) | 26.78 (2.690) | 25.90 (3.502) | 27.02 (3.609) | 27.29 (3.311) | 27.11 (3.740) | 28.64 (2.978) | 27.78 (2.606) | 26.05 (3.345) | 27.02 (3.163)
Body Mass Index [Median (Full Range); unit: kg/m^2] | 27.95 [22.2 to 30.9] | 26.95 [22.4 to 29.8] | 25.20 [21.6 to 31.3] | 28.70 [20.0 to 30.8] | 27.30 [23.3 to 31.2] | 27.00 [19.7 to 31.7] | 29.35 [23.8 to 31.8] | 26.80 [24.6 to 31.7] | 26.05 [21.1 to 30.5] | 27.00 [19.7 to 31.8]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) After a Single Dose of CD388
Description: Number of participants with at least one TEAE, including but not limited to adverse events (AEs) and serious adverse events (SAEs) (including systemic reactogenicity/injection site reactions and hypersensitivity reactions), and AEs leading to study drug discontinuation and/or study withdrawal, based on vital signs, 12-lead electrocardiogram (ECG), and clinical laboratory test (hematology, coagulation, serum chemistry, and urinalysis) abnormalities following a single dose of CD388.
Time Frame: Day 1 through Day 120 (±14 days; Cohorts 1A/1B only); Day 1 through Day 374 (±14 days; Cohorts 2A/2B and 3A/3B); or Day 1 through Day 206 (±10 days; Cohort 4B only)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- CD388 50 mg IM: Participants randomized to Cohort 1A to receive a single dose of 50 milligrams (mg) CD388, administered by intramuscular (IM) injection.
  CD388: CD388 liquid for injection
- CD388 150 mg IM: Participants randomized to Cohort 2A to receive a single dose of 150 mg CD388, administered by IM injection, followed by another single dose of the same treatment administered by the same route after washout of 5 effective half-lives after the first dose.
  CD388: CD388 liquid for injection
- CD388 450 mg IM: Participants randomized to Cohort 3A to receive a single dose of 450 mg CD388, administered by IM injection, followed by another single dose of the same treatment administered by the same route after washout of 5 effective half-lives after the first dose.
  CD388: CD388 liquid for injection
- Pooled Placebo IM: Participants randomized to Cohort 1A, 2A, or 3A to receive a single dose of saline placebo, administered by IM injection. Of these participants, those that advanced through the study in cohorts with participants in the CD388 150 mg IM (Cohort 2A) and CD388 450 mg IM (Cohort 3A) arms received another single dose of saline placebo administered by the same route after washout of 5 effective half-lives after the first dose.
  Saline placebo: Sterile normal saline for injection
- CD388 50 mg SQ: Participants randomized to Cohort 1B to receive a single dose of 50 mg CD388, administered by subcutaneous (SQ) injection.
  CD388: CD388 liquid for injection
- CD388 150 mg SQ: Participants randomized to Cohort 2B to receive a single dose of 150 mg CD388, administered by SQ injection, followed by another single dose of the same treatment administered by the same route after washout of 5 effective half-lives after the first dose.
  CD388: CD388 liquid for injection
- CD388 450 mg SQ: Participants randomized to Cohort 3B to receive a single dose of 450 mg CD388, administered by SQ injection, followed by another single dose of the same treatment administered by the same route after washout of 5 effective half-lives after the first dose.
  CD388: CD388 liquid for injection
- CD388 900 mg SQ: Participants randomized to Cohort 4B to receive a single dose of 900 mg CD388, administered by SQ injection.
  CD388: CD388 liquid for injection
- Pooled Placebo SQ: Participants randomized to Cohort 1B, 2B, 3B, or 4B to receive a single dose of saline placebo, administered by SQ injection. Of these participants, those that advanced through the study in cohorts with participants in the CD388 150 mg SQ (Cohort 2B) and CD388 450 mg SQ (Cohort 3B) arms received another single dose of saline placebo administered by the same route after washout of 5 effective half-lives after the first dose.
  Saline placebo: Sterile normal saline for injection
Arm/Group | CD388 50 mg IM | CD388 150 mg IM | CD388 450 mg IM | Pooled Placebo IM | CD388 50 mg SQ | CD388 150 mg SQ | CD388 450 mg SQ | CD388 900 mg SQ | Pooled Placebo SQ
Number analyzed (Participants) | 8 | 8 | 8 | 9 | 8 | 8 | 8 | 8 | 12
Participants
  Participants with at least one TEAE | 5 | 5 | 5 | 8 | 5 | 4 | 5 | 3 | 7
  Participants with AEs leading to study withdrawal | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0

2. Primary Outcome: Severity of TEAEs After a Single Dose of CD388
Description: Maximum severity of TEAEs reported (in participants with at least one TEAE), including but not limited to adverse events (AEs) and serious adverse events (SAEs) (including systemic reactogenicity/injection site reactions and hypersensitivity reactions), and AEs leading to study drug discontinuation and/or study withdrawal, based on vital signs, electrocardiogram (ECG), and clinical laboratory test (including hematology, coagulation, serum chemistry, and urinalysis) abnormalities following a single dose of CD388.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | CD388 50 mg IM | CD388 150 mg IM | CD388 450 mg IM | Pooled Placebo IM | CD388 50 mg SQ | CD388 150 mg SQ | CD388 450 mg SQ | CD388 900 mg SQ | Pooled Placebo SQ
Number analyzed (Participants) | 8 | 8 | 8 | 9 | 8 | 8 | 8 | 8 | 12
Participants
  Mild | 5 | 5 | 2 | 5 | 4 | 4 | 3 | 3 | 6
  Moderate | 0 | 0 | 3 | 2 | 1 | 0 | 1 | 0 | 1
  Severe | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0

3. Secondary Outcome: Mean Peak Plasma Concentration (Cmax) Following a Single Administration of CD388
Description: Evaluation of the maximum plasma concentration (Cmax) following the first single dose of CD388 administered by either IM or SQ injection.
Time Frame: Days 1 through 7, 9, 11, 14, 21, and 30 (all cohorts) and at outpatient visits: Days 45, 60, 90, and 120 (Cohorts 1A/1B only); Days 45, 84, 126, and 168 (Cohorts 2A/2B and 3A/3B); or Days 45, 84, 126, 168, and 206 (Cohort 4B only)
Population: The Pharmacokinetic (PK) Population included all randomized participants who received at least a portion of 1 dose of CD388 and had at least 1 evaluable post-dose concentration value. Participants administered matching placebo were not included in the PK Population.
Measure: Mean (Standard Deviation); unit: micrograms/milliliter (ug/mL)
Groups:
- Cohort 1A CD388 50 mg IM: Participants randomized to receive a single dose of 50 milligrams (mg) CD388, administered by intramuscular (IM) injection.
- Cohort 2A CD388 150 mg IM: Participants randomized to receive a single dose of 150 mg CD388, administered by IM injection, followed by another single dose of the same treatment administered by the same route after washout of 5 effective half-lives after the first dose.
- Cohort 3A CD388 450 mg IM: Participants randomized to receive a single dose of 450 mg CD388, administered by IM injection, followed by another single dose of the same treatment administered by the same route after washout of 5 effective half-lives after the first dose.
- Cohort 1B CD388 50 mg SQ: Participants randomized to receive a single dose of 50 mg CD388, administered by subcutaneous (SQ) injection.
- Cohort 2B CD388 150 mg SQ: Participants randomized to receive a single dose of 150 mg CD388, administered by SQ injection, followed by another single dose of the same treatment administered by the same route after washout of 5 effective half-lives after the first dose.
- Cohort 3B CD388 450 mg SQ: Participants randomized to receive a single dose of 450 mg CD388, administered by SQ injection, followed by another single dose of the same treatment administered by the same route after washout of 5 effective half-lives after the first dose.
- Cohort 4B CD388 900 mg SQ: Participants randomized to receive a single dose of 900 mg CD388, administered by SQ injection.
Arm/Group | Cohort 1A CD388 50 mg IM | Cohort 2A CD388 150 mg IM | Cohort 3A CD388 450 mg IM | Cohort 1B CD388 50 mg SQ | Cohort 2B CD388 150 mg SQ | Cohort 3B CD388 450 mg SQ | Cohort 4B CD388 900 mg SQ
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8
micrograms/milliliter (ug/mL) | 4.13 (0.747) | 10.4 (2.44) | 48.6 (11.7) | 3.57 (0.942) | 12.0 (3.35) | 32.7 (9.40) | 58.8 (17.5)

4. Secondary Outcome: Median Peak Plasma Concentration (Cmax) Following a Single Administration of CD388
Description: as for outcome 3
Time Frame: as for outcome 3
Population: The PK Population included all randomized participants who received at least a portion of 1 dose of CD388 and had at least 1 evaluable post-dose concentration value. Participants administered matching placebo were not included in the PK Population.
Measure: Median (Full Range); unit: micrograms/milliliter (ug/mL)
Arm/Group | Cohort 1A CD388 50 mg IM | Cohort 2A CD388 150 mg IM | Cohort 3A CD388 450 mg IM | Cohort 1B CD388 50 mg SQ | Cohort 2B CD388 150 mg SQ | Cohort 3B CD388 450 mg SQ | Cohort 4B CD388 900 mg SQ
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8
micrograms/milliliter (ug/mL) | 3.96 [2.91 to 5.34] | 10.4 [6.52 to 13.6] | 48.0 [35.2 to 67.7] | 3.72 [2.17 to 4.83] | 11.8 [6.84 to 17.0] | 31.6 [16.6 to 48.0] | 60.7 [34.3 to 91.3]

5. Secondary Outcome: Mean Time to Maximum Plasma Concentration (Tmax) Following a Single Administration of CD388
Description: Evaluation of the time to maximum plasma concentration (Tmax) following the first single dose of CD388 administered by either IM or SQ injection.
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hours (h)
Arm/Group | Cohort 1A CD388 50 mg IM | Cohort 2A CD388 150 mg IM | Cohort 3A CD388 450 mg IM | Cohort 1B CD388 50 mg SQ | Cohort 2B CD388 150 mg SQ | Cohort 3B CD388 450 mg SQ | Cohort 4B CD388 900 mg SQ
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8
hours (h) | 111.08 (72.42) | 159.03 (83.10) | 85.64 (42.19) | 213.00 (108.43) | 137.48 (77.82) | 120.04 (67.83) | 109.54 (55.66)

6. Secondary Outcome: Median Time to Maximum Plasma Concentration (Tmax) Following a Single Administration of CD388
Description: as for outcome 5
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Cohort 1A CD388 50 mg IM | Cohort 2A CD388 150 mg IM | Cohort 3A CD388 450 mg IM | Cohort 1B CD388 50 mg SQ | Cohort 2B CD388 150 mg SQ | Cohort 3B CD388 450 mg SQ | Cohort 4B CD388 900 mg SQ
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8
hours (h) | 96.07 [48.17 to 240.00] | 131.98 [71.97 to 312.00] | 78.31 [24.17 to 144.00] | 228.00 [72.00 to 312.02] | 131.28 [48.22 to 312.02] | 96.00 [48.17 to 240.00] | 96.00 [48.17 to 192.00]

7. Secondary Outcome: Mean Terminal Elimination Half-life (t½) Following a Single Administration of CD388
Description: Evaluation of the terminal elimination half-life (t½) following the first single dose of CD388 administered by either IM or SQ injection.
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hours (h)
Arm/Group | Cohort 1A CD388 50 mg IM | Cohort 2A CD388 150 mg IM | Cohort 3A CD388 450 mg IM | Cohort 1B CD388 50 mg SQ | Cohort 2B CD388 150 mg SQ | Cohort 3B CD388 450 mg SQ | Cohort 4B CD388 900 mg SQ
Number analyzed (Participants) | 8 | 7 | 8 | 8 | 8 | 8 | 8
hours (h) | 1234.41 (140.04) | 1192.03 (235.80) | 1006.20 (314.39) | 1069.78 (216.48) | 1265.53 (223.93) | 1065.21 (239.19) | 1384.36 (282.53)

8. Secondary Outcome: MedianTerminal Elimination Half-life (t½) Following a Single Administration of CD388
Description: as for outcome 7
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Cohort 1A CD388 50 mg IM | Cohort 2A CD388 150 mg IM | Cohort 3A CD388 450 mg IM | Cohort 1B CD388 50 mg SQ | Cohort 2B CD388 150 mg SQ | Cohort 3B CD388 450 mg SQ | Cohort 4B CD388 900 mg SQ
Number analyzed (Participants) | 8 | 7 | 8 | 8 | 8 | 8 | 8
hours (h) | 1275.62 [985.09 to 1390.45] | 1285.85 [783.24 to 1471.71] | 1137.42 [540.88 to 1384.09] | 1052.39 [685.81 to 1350.50] | 1270.40 [796.65 to 1576.21] | 1040.30 [809.64 to 1502.38] | 1287.45 [1110.87 to 1998.04]

9. Secondary Outcome: Mean Apparent Clearance (CL/F) Following a Single Administration of CD388
Description: Evaluation of the apparent clearance (CL/F) following the first single dose of CD388 administered by either IM or SQ injection.
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: liters/hour (L/h)
Arm/Group | Cohort 1A CD388 50 mg IM | Cohort 2A CD388 150 mg IM | Cohort 3A CD388 450 mg IM | Cohort 1B CD388 50 mg SQ | Cohort 2B CD388 150 mg SQ | Cohort 3B CD388 450 mg SQ | Cohort 4B CD388 900 mg SQ
Number analyzed (Participants) | 8 | 7 | 8 | 8 | 8 | 8 | 8
liters/hour (L/h) | 0.00751 (0.00119) | 0.00867 (0.00177) | 0.00766 (0.00199) | 0.00900 (0.00230) | 0.00725 (0.00123) | 0.00883 (0.00213) | 0.00863 (0.00158)

10. Secondary Outcome: Median Apparent Clearance (CL/F) Following a Single Administration of CD388
Description: as for outcome 9
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Median (Full Range); unit: liters/hour (L/h)
Arm/Group | Cohort 1A CD388 50 mg IM | Cohort 2A CD388 150 mg IM | Cohort 3A CD388 450 mg IM | Cohort 1B CD388 50 mg SQ | Cohort 2B CD388 150 mg SQ | Cohort 3B CD388 450 mg SQ | Cohort 4B CD388 900 mg SQ
Number analyzed (Participants) | 8 | 7 | 8 | 8 | 8 | 8 | 8
liters/hour (L/h) | 0.00707 [0.00614 to 0.00991] | 0.00851 [0.00640 to 0.0112] | 0.00726 [0.00571 to 0.0116] | 0.00834 [0.00591 to 0.0128] | 0.00717 [0.00551 to 0.00909] | 0.00912 [0.00493 to 0.0115] | 0.00870 [0.00648 to 0.0111]

11. Secondary Outcome: Mean Apparent Volume of Distribution (V[z]/F) Following a Single Administration of CD388
Description: Evaluation of the apparent volume of distribution (V[z]/F) following the first single dose of CD388 administered by either IM or SQ injection.
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: liters (L)
Arm/Group | Cohort 1A CD388 50 mg IM | Cohort 2A CD388 150 mg IM | Cohort 3A CD388 450 mg IM | Cohort 1B CD388 50 mg SQ | Cohort 2B CD388 150 mg SQ | Cohort 3B CD388 450 mg SQ | Cohort 4B CD388 900 mg SQ
Number analyzed (Participants) | 8 | 7 | 8 | 8 | 8 | 8 | 8
liters (L) | 13.3 (1.91) | 14.8 (4.40) | 10.7 (2.99) | 13.4 (2.59) | 13.3 (3.70) | 13.1 (2.61) | 17.1 (3.76)

12. Secondary Outcome: Median Apparent Volume of Distribution (V[z]/F) Following a Single Administration of CD388
Description: as for outcome 11
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Median (Full Range); unit: liters (L)
Arm/Group | Cohort 1A CD388 50 mg IM | Cohort 2A CD388 150 mg IM | Cohort 3A CD388 450 mg IM | Cohort 1B CD388 50 mg SQ | Cohort 2B CD388 150 mg SQ | Cohort 3B CD388 450 mg SQ | Cohort 4B CD388 900 mg SQ
Number analyzed (Participants) | 8 | 7 | 8 | 8 | 8 | 8 | 8
liters (L) | 13.9 [10.3 to 15.8] | 14.4 [11.1 to 23.9] | 10.9 [6.47 to 15.1] | 12.2 [11.4 to 18.7] | 12.7 [9.27 to 20.7] | 12.9 [10.7 to 18.9] | 16.7 [11.2 to 24.2]

13. Secondary Outcome: Mean Area Under the Plasma Concentration-Time Curve From Time 0 to Time of Last Quantifiable Sample (AUC[0-t]) Following a Single Administration of CD388
Description: Evaluation of the area under the plasma concentration-time curve from time 0 to time of last quantifiable sample (AUC[0-t]) following the first single dose of CD388 administered by either IM or SQ injection.
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ug*h/mL
Arm/Group | Cohort 1A CD388 50 mg IM | Cohort 2A CD388 150 mg IM | Cohort 3A CD388 450 mg IM | Cohort 1B CD388 50 mg SQ | Cohort 2B CD388 150 mg SQ | Cohort 3B CD388 450 mg SQ | Cohort 4B CD388 900 mg SQ
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8
ug*h/mL | 5450 (728) | 15000 (4320) | 53800 (12000) | 4830 (965) | 18800 (3360) | 49000 (13100) | 96300 (16700)

14. Secondary Outcome: Median Area Under the Plasma Concentration-Time Curve From Time 0 to Time of Last Quantifiable Sample (AUC[0-t]) Following a Single Administration of CD388
Description: as for outcome 13
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Median (Full Range); unit: ug*h/mL
Arm/Group | Cohort 1A CD388 50 mg IM | Cohort 2A CD388 150 mg IM | Cohort 3A CD388 450 mg IM | Cohort 1B CD388 50 mg SQ | Cohort 2B CD388 150 mg SQ | Cohort 3B CD388 450 mg SQ | Cohort 4B CD388 900 mg SQ
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8
ug*h/mL | 5460 [4410 to 6530] | 15100 [7250 to 21100] | 52100 [37600 to 71200] | 4960 [3270 to 6300] | 18700 [13700 to 24400] | 46500 [34800 to 76600] | 94700 [71700 to 121000]

15. Secondary Outcome: Mean Area Under the Plasma Concentration-Time Curve From Time 0 Extrapolated to Infinity (AUC[0-∞]) Following a Single Administration of CD388
Description: Evaluation of the area under the plasma concentration-time curve from time 0 extrapolated to infinity (AUC[0-∞]) following the first single dose of CD388 administered by either IM or SQ injection.
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ug*h/mL
Arm/Group | Cohort 1A CD388 50 mg IM | Cohort 2A CD388 150 mg IM | Cohort 3A CD388 450 mg IM | Cohort 1B CD388 50 mg SQ | Cohort 2B CD388 150 mg SQ | Cohort 3B CD388 450 mg SQ | Cohort 4B CD388 900 mg SQ
Number analyzed (Participants) | 8 | 7 | 8 | 8 | 8 | 8 | 8
ug*h/mL | 6790 (973) | 17900 (3670) | 61800 (13600) | 5870 (1470) | 21200 (3670) | 54400 (16900) | 107000 (19700)

16. Secondary Outcome: Median Area Under the Plasma Concentration-Time Curve From Time 0 Extrapolated to Infinity (AUC[0-∞]) Following a Single Administration of CD388
Description: as for outcome 15
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Median (Full Range); unit: ug*h/mL
Arm/Group | Cohort 1A CD388 50 mg IM | Cohort 2A CD388 150 mg IM | Cohort 3A CD388 450 mg IM | Cohort 1B CD388 50 mg SQ | Cohort 2B CD388 150 mg SQ | Cohort 3B CD388 450 mg SQ | Cohort 4B CD388 900 mg SQ
Number analyzed (Participants) | 8 | 7 | 8 | 8 | 8 | 8 | 8
ug*h/mL | 7080 [5050 to 8140] | 17600 [13300 to 23400] | 62100 [38800 to 78800] | 6000 [3920 to 8470] | 21000 [16500 to 27200] | 49300 [39100 to 91400] | 103000 [80800 to 139000]

17. Secondary Outcome: Mean Peak Plasma Concentration (Cmax) Following a Repeated Single Administration of CD388
Description: Evaluation of the maximum plasma concentration (Cmax) following a repeated single dose of CD388 administered by either IM or SQ injection (after washout of 5 effective half-lives from the first dose).
Time Frame: At inpatient visits on Days 206 (i.e., Dose 2 Day 1) through 212, 214, 216, 219, 226, and 236; and at outpatient visits: Days 251, 290, 332, and 374 (Cohorts 2A/2B and 3A/3B only)
Population: The PK Completer Population included all randomized participants who received 2 single doses of CD388 and obtained adequate PK samples for PK parameter estimation. Participants administered matching placebo were not included in the Completer PK Population.
Measure: Mean (Standard Deviation); unit: micrograms/milliliter (ug/mL)
Arm/Group | Cohort 2A CD388 150 mg IM | Cohort 3A CD388 450 mg IM | Cohort 2B CD388 150 mg SQ | Cohort 3B CD388 450 mg SQ
Number analyzed (Participants) | 6 | 7 | 8 | 5
micrograms/milliliter (ug/mL) | 10.5 (3.30) | 28.8 (7.66) | 13.0 (5.34) | 31.1 (7.86)

18. Secondary Outcome: Median Peak Plasma Concentration (Cmax) Following a Repeated Single Administration of CD388
Description: as for outcome 17
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Median (Full Range); unit: micrograms/milliliter (ug/mL)
Arm/Group | Cohort 2A CD388 150 mg IM | Cohort 3A CD388 450 mg IM | Cohort 2B CD388 150 mg SQ | Cohort 3B CD388 450 mg SQ
Number analyzed (Participants) | 6 | 7 | 8 | 5
micrograms/milliliter (ug/mL) | 9.94 [6.68 to 14.4] | 29.8 [18.0 to 38.3] | 12.5 [6.84 to 22.0] | 29.3 [23.8 to 43.8]

19. Secondary Outcome: Mean Time to Maximum Plasma Concentration (Tmax) Following a Repeated Single Administration of CD388
Description: Evaluation of the time to maximum plasma concentration (Tmax) following a repeated single dose of CD388 administered by either IM or SQ injection (after washout of 5 effective half-lives from the first dose).
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: hours (h)
Arm/Group | Cohort 2A CD388 150 mg IM | Cohort 3A CD388 450 mg IM | Cohort 2B CD388 150 mg SQ | Cohort 3B CD388 450 mg SQ
Number analyzed (Participants) | 6 | 7 | 8 | 5
hours (h) | 104.02 (81.25) | 161.14 (75.53) | 251.99 (200.79) | 105.02 (49.89)

20. Secondary Outcome: Median Time to Maximum Plasma Concentration (Tmax) Following a Repeated Single Administration of CD388
Description: as for outcome 19
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Cohort 2A CD388 150 mg IM | Cohort 3A CD388 450 mg IM | Cohort 2B CD388 150 mg SQ | Cohort 3B CD388 450 mg SQ
Number analyzed (Participants) | 6 | 7 | 8 | 5
hours (h) | 84.00 [48.00 to 264.00] | 144.00 [48.00 to 264.00] | 227.99 [48.00 to 695.97] | 96.00 [47.07 to 167.00]

21. Secondary Outcome: Mean Terminal Elimination Half-life (t½) Following a Repeated Single Administration of CD388
Description: Evaluation of the terminal elimination half-life (t½) following a repeated single dose of CD388 administered by either IM or SQ injection (after washout of 5 effective half-lives from the first dose).
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: hours (h)
Arm/Group | Cohort 2A CD388 150 mg IM | Cohort 3A CD388 450 mg IM | Cohort 2B CD388 150 mg SQ | Cohort 3B CD388 450 mg SQ
Number analyzed (Participants) | 6 | 7 | 8 | 5
hours (h) | 1324.07 (198.33) | 1408.43 (336.72) | 1059.55 (409.51) | 1301.42 (83.00)

22. Secondary Outcome: Median Terminal Elimination Half-life (t½) Following a Repeated Single Administration of CD388
Description: as for outcome 21
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Cohort 2A CD388 150 mg IM | Cohort 3A CD388 450 mg IM | Cohort 2B CD388 150 mg SQ | Cohort 3B CD388 450 mg SQ
Number analyzed (Participants) | 6 | 7 | 8 | 5
hours (h) | 1342.81 [1108.91 to 1639.43] | 1506.38 [670.64 to 1721.28] | 1218.60 [508.57 to 1539.09] | 1348.40 [1175.81 to 1371.62]

23. Secondary Outcome: Mean Apparent Clearance (CL/F) Following a Repeated Single Administration of CD388
Description: Evaluation of the apparent clearance (CL/F) following a repeated single dose of CD388 administered by either IM or SQ injection (after washout of 5 effective half-lives from the first dose).
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: liters/hour (L/h)
Arm/Group | Cohort 2A CD388 150 mg IM | Cohort 3A CD388 450 mg IM | Cohort 2B CD388 150 mg SQ | Cohort 3B CD388 450 mg SQ
Number analyzed (Participants) | 6 | 7 | 8 | 5
liters/hour (L/h) | 0.00923 (0.00123) | 0.00886 (0.00170) | 0.00802 (0.00218) | 0.00897 (0.00210)

24. Secondary Outcome: Median Apparent Clearance (CL/F) Following a Repeated Single Administration of CD388
Description: as for outcome 23
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Median (Full Range); unit: liters/hour (L/h)
Arm/Group | Cohort 2A CD388 150 mg IM | Cohort 3A CD388 450 mg IM | Cohort 2B CD388 150 mg SQ | Cohort 3B CD388 450 mg SQ
Number analyzed (Participants) | 6 | 7 | 8 | 5
liters/hour (L/h) | 0.00954 [0.00706 to 0.0104] | 0.00918 [0.00642 to 0.0105] | 0.00866 [0.00507 to 0.0116] | 0.00946 [0.00534 to 0.0106]

25. Secondary Outcome: Mean Apparent Volume of Distribution (V[z]/F) Following a Repeated Single Administration of CD388
Description: Evaluation of the apparent volume of distribution (V[z]/F) following a repeated single dose of CD388 administered by either IM or SQ injection (after washout of 5 effective half-lives from the first dose).
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: liters (L)
Arm/Group | Cohort 2A CD388 150 mg IM | Cohort 3A CD388 450 mg IM | Cohort 2B CD388 150 mg SQ | Cohort 3B CD388 450 mg SQ
Number analyzed (Participants) | 6 | 7 | 8 | 5
liters (L) | 17.4 (1.85) | 17.8 (5.45) | 11.7 (4.70) | 16.7 (3.55)

26. Secondary Outcome: Median Apparent Volume of Distribution (V[z]/F) Following a Repeated Single Administration of CD388
Description: as for outcome 25
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Median (Full Range); unit: liters (L)
Arm/Group | Cohort 2A CD388 150 mg IM | Cohort 3A CD388 450 mg IM | Cohort 2B CD388 150 mg SQ | Cohort 3B CD388 450 mg SQ
Number analyzed (Participants) | 6 | 7 | 8 | 5
liters (L) | 16.6 [15.4 to 20.2] | 16.7 [10.1 to 26.0] | 9.46 [7.45 to 19.2] | 18.3 [10.4 to 18.5]

27. Secondary Outcome: Mean Area Under the Plasma Concentration-Time Curve From Time 0 to Time of Last Quantifiable Sample (AUC[0-t]) Following a Repeated Single Administration of CD388
Description: Evaluation of the area under the plasma concentration-time curve from time 0 to time of last quantifiable sample (AUC[0-t]) following a repeated single dose of CD388 administered by either IM or SQ injection (after washout of 5 effective half-lives from the first dose).
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ug*h/mL
Arm/Group | Cohort 2A CD388 150 mg IM | Cohort 3A CD388 450 mg IM | Cohort 2B CD388 150 mg SQ | Cohort 3B CD388 450 mg SQ
Number analyzed (Participants) | 6 | 7 | 8 | 5
ug*h/mL | 14400 (2050) | 41300 (15400) | 18000 (5090) | 41100 (21100)

28. Secondary Outcome: Median Area Under the Plasma Concentration-Time Curve From Time 0 to Time of Last Quantifiable Sample (AUC[0-t]) Following a Repeated Single Administration of CD388
Description: as for outcome 27
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Median (Full Range); unit: ug*h/mL
Arm/Group | Cohort 2A CD388 150 mg IM | Cohort 3A CD388 450 mg IM | Cohort 2B CD388 150 mg SQ | Cohort 3B CD388 450 mg SQ
Number analyzed (Participants) | 6 | 7 | 8 | 5
ug*h/mL | 13600 [12800 to 18000] | 41800 [13400 to 60600] | 16000 [12900 to 26600] | 39100 [13400 to 72700]

29. Secondary Outcome: Mean Area Under the Plasma Concentration-Time Curve From Time 0 Extrapolated to Infinity (AUC[0-∞]) Following a Repeated Single Administration of CD388
Description: Evaluation of the area under the plasma concentration-time curve from time 0 extrapolated to infinity (AUC[0-∞]) following a repeated single dose of CD388 administered by either IM or SQ injection (after washout of 5 effective half-lives from the first dose).
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ug*h/mL
Arm/Group | Cohort 2A CD388 150 mg IM | Cohort 3A CD388 450 mg IM | Cohort 2B CD388 150 mg SQ | Cohort 3B CD388 450 mg SQ
Number analyzed (Participants) | 6 | 7 | 8 | 5
ug*h/mL | 16500 (2530) | 52600 (10800) | 20000 (5830) | 53400 (17400)

30. Secondary Outcome: Median Area Under the Plasma Concentration-Time Curve From Time 0 Extrapolated to Infinity (AUC[0-∞]) Following a Repeated Single Administration of CD388
Description: as for outcome 29
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Median (Full Range); unit: ug*h/mL
Arm/Group | Cohort 2A CD388 150 mg IM | Cohort 3A CD388 450 mg IM | Cohort 2B CD388 150 mg SQ | Cohort 3B CD388 450 mg SQ
Number analyzed (Participants) | 6 | 7 | 8 | 5
ug*h/mL | 15700 [14500 to 21200] | 49000 [42900 to 70100] | 17300 [12900 to 29600] | 47600 [42300 to 84300]

31. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) After a Repeated Single Dose of CD388
Description: Number of participants with at least one TEAE, including but not limited to AEs and SAEs (including systemic reactogenicity/injection site reactions and hypersensitivity reactions), and AEs leading to study drug discontinuation and/or study withdrawal, based on vital signs, 12-lead ECG, and clinical laboratory test (hematology, coagulation, serum chemistry, and urinalysis) abnormalities following a repeated single dose of CD388.
Time Frame: Day 207 through Day 412 (±10 days) (Cohorts 2A/2B and 3A/3B only)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Pooled Placebo IM: Participants randomized to Cohort 2A or 3A to receive a single dose of saline placebo, administered by IM injection, followed by another single dose of the same treatment administered by the same route after washout of 5 effective half-lives after the first dose.
  Saline placebo: Sterile normal saline for injection
- Pooled Placebo SQ: Participants randomized to Cohort 2B or 3B to receive a single dose of saline placebo, administered by SQ injection, followed by another single dose of the same treatment administered by the same route after washout of 5 effective half-lives after the first dose.
  Saline placebo: Sterile normal saline for injection
Arm/Group | CD388 150 mg IM | CD388 450 mg IM | Pooled Placebo IM | CD388 150 mg SQ | CD388 450 mg SQ | Pooled Placebo SQ
Number analyzed (Participants) | 6 | 7 | 4 | 8 | 5 | 4
Participants
  Participants with at least one TEAE | 2 | 4 | 2 | 2 | 3 | 1
  Participants with AEs leading to study withdrawal | 0 | 0 | 0 | 0 | 0 | 0

32. Secondary Outcome: Severity of TEAEs After a Repeated Single Dose of CD388
Description: Maximum severity of TEAEs reported (in participants with at least one TEAE), including but not limited to AEs and SAEs (including systemic reactogenicity/injection site reactions and hypersensitivity reactions), and AEs leading to study drug discontinuation and/or study withdrawal, based on vital signs, 12-lead ECG, and clinical laboratory test (including hematology, coagulation, serum chemistry, and urinalysis) abnormalities following a repeated single dose of CD388.
Time Frame: Day 207 through Day 412 (±10 days) (Cohorts 2A/2B and 3A/3B only)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | CD388 150 mg IM | CD388 450 mg IM | Pooled Placebo IM | CD388 150 mg SQ | CD388 450 mg SQ | Pooled Placebo SQ
Number analyzed (Participants) | 6 | 7 | 4 | 8 | 5 | 4
Participants
  Mild | 2 | 2 | 2 | 2 | 3 | 1
  Moderate | 0 | 2 | 0 | 0 | 0 | 0
  Severe | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for all participants from the time of signing the informed consent form through the final study visit (Day 120 for the 50 mg dose arm [Cohorts 1A/1B]; Day 412 for the 150 mg and 450 mg dose arms [Cohorts 2A/2B and 3A/3B]; and Day 206 for the 900 mg dose arm [Cohort 4B]).
Description: All-Cause Mortality, Serious Adverse Events, and Other (Not Including Serious) Adverse Events were assessed in the Safety Population, which included all randomized participants who received any amount of study drug (77 total; 33 [IM route], 44 [SQ route]).
Arm/Group | CD388 50 mg IM | CD388 150 mg IM | CD388 450 mg IM | Pooled Placebo IM | CD388 50 mg SQ | CD388 150 mg SQ | CD388 450 mg SQ | CD388 900 mg SQ | Pooled Placebo SQ
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/9 | 0/8 | 0/8 | 0/8 | 0/8 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/9 | 0/8 | 0/8 | 0/8 | 0/8 | 0/12
Other Adverse Events (participants affected / at risk) | 5/8 | 5/8 | 6/8 | 8/9 | 5/8 | 4/8 | 6/8 | 3/8 | 7/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CD388 50 mg IM (N=8) | CD388 150 mg IM (N=8) | CD388 450 mg IM (N=8) | Pooled Placebo IM (N=9) | CD388 50 mg SQ (N=8) | CD388 150 mg SQ (N=8) | CD388 450 mg SQ (N=8) | CD388 900 mg SQ (N=8) | Pooled Placebo SQ (N=12)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Saliva discoloration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (3) | 2 (4) | 4 (8) | 5 (10) | 0 (0) | 2 (4) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Feces hard (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (2) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
COVID-19 (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pustule (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site hemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site hematoma (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure systolic increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure diastolic increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital edema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post inflammatory pigmentation change (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic hematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nodal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2023-02-07): https://cdn.clinicaltrials.gov/large-docs/37/NCT05285137/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/37/NCT05285137/SAP_001.pdf